CLINICAL TRIAL: NCT01120015
Title: Phase 4 Study of Diacerein as Adjuvant to Diclofenac Sodium in Indian Patients of OA Knee
Brief Title: Diacerein as Adjuvant to Diclofenac Sodium in Indian Patients of Osteoarthritis (OA) Knee
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Government Medical College, Amritsar (Other Government)
Responsible Party: Kuljinder singh, Pharmacology department
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ks1
Record Dates: First submitted 2010-05-07; First posted 2010-05-10 (Estimated); Last update posted 2010-05-31 (Estimated); Status verified 2009-05

CONDITIONS: Osteoarthritis; Osteoarthritis, Knee
Keywords: OA; knee
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee | interventions — diacerein

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diacerein (Experimental): diacerein 50mg oD first month, 50 mg BD next 2 months
  Interventions: Drug: diacerein

INTERVENTIONS:
Drug: diacerein — Diclofenac sodium 75mg sustained release tablet once daily was given to both groups for 3 months. Capsule diacerein 50mg in study group and matched placebo in control group were given once daily for first month and twice daily for next two months with the main meals.

SUMMARY:
The purpose of this study is to evaluate clinical effectiveness of diacerein as add on therapy to diclofenac sodium in Indian patients of osteoarthritis (OA) knee.

DETAILED DESCRIPTION:
Currently symptomatic relief is provided by the use of nonsteroidal anti-inflammatory drugs (NSAIDs) but they do not reverse the basic pathology of disease, rather may accelerate it, like degeneration of cartilage, inhibition of chondroitin synthesis and suppression of proteoglycans synthesis by the chondrocyte.

Research shows that IL-1β plays a fundamental role in osteoarthritis pathophysiology and cartilage destruction. Diacerein, a purified compound with anthraquinonic structure, inhibits IL-1β, retarding all pathological processes initiated in OA. Also, Diacerein has proven analgesic efficacy comparable to that of diclofenac in patients of osteoarthritis knee12. Because of these factors, the present study has been planned to evaluate the clinical effectiveness of diacerein as add on therapy to diclofenac sodium in Indian patients of symptomatic OA knee.

ELIGIBILITY:
Inclusion Criteria:

* Primary osteoarthritis Patients recruited were between 35 to 60 years of age, with X-ray confirmed Kellgren-Lawrence grade13 II or III severity primary tibiofemoral OA, according to the American College of Rheumatology criteria.
* Women of childbearing age had to provide evidence of adequate contraception prior to inclusion.

Exclusion Criteria:

Those patients were excluded from the present study who:

* were of age less than 35 years or more than 60 years
* presented with active concomitant gastroduodenal disorders, hepatic and renal impairment within last 30 days prior to receiving the study drug
* were diagnosed to have any inflammatory arthritis, gout or acute trauma of the knee, hip or spine; accompanying OA of the hip of sufficient severity to interfere with the functional assessment of the knee
* had previous or ongoing treatment with oral SYSDOA (e.g., glucosamine sulphate, chondroitin sulphate, diacerein, piascledine), anti-depressants, tranquillisers, antacids or antibiotics; were having active cardiac lesion or hypertension, were pregnant females and those who were planning their pregnancy during the study
* were having a known hypersensitivity to diclofenac sodium, to diacerein, to similar compounds, to the excipients or paracetamol, have history of painful knee conditions other than OA
* have persistent diarrhoea or laxative use; severe gastrointestinal disorders, severe obesity, severe parenchymal organ disease, or anaemia (haemoglobin< 10.0 g/ dl or haematocrit < 30%).
* Patients who received oral, intramuscular, intraarticular or soft tissue injections of corticosteroids within last eight weeks before receiving the first dose of the study medication, or had undergone joint lavage and arthroscopic procedures in the previous 6 months, were also excluded.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2007-01; Primary Completion 2008-06 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Visual Analogue scale assessment of pain .

SECONDARY OUTCOMES:
WOMAC assessment of pain, physical function
Global patient and physician assessment of pain and function
Paracetamol consumption

CONTACTS AND LOCATIONS:
Overall Officials: Kuljinder Singh, MD, Principal Investigator — GMC Amritsar; Jaswant rai, MD, Study Chair — GMC Amritsar; Rakesh sharma, MS, Study Chair — GMC Amritsar
Locations (1):
- Kuljinder Singh, Amritsar, Punjab, India